CLINICAL TRIAL: NCT07049380
Title: Post-Operative Analgesic Effect of Tramadol and Nalbuphine in Smoker and Non-Smoker Patients Following Laparoscopic Cholecystectomy
Brief Title: Post-Operative Analgesic Effect of Tramadol and Nalbuphine in Smoker and Non-Smoker Patients in LC
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/910
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Laparocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comparative cross sectional — evaluating the efficacy of two analgesics, tramadol and nalbuphine. The primary objectives are to estimate pain severity in smokers versus nonsmokers and identify the effect of tramadol and nalbuphine between these groups

SUMMARY:
This study aims to compare pain severity and analgesic requirements between smokers and nonsmokers following laparoscopic cholecystectomy, evaluating the efficacy of two analgesics, tramadol and nalbuphine.

DETAILED DESCRIPTION:
The primary objectives are to estimate pain severity in smokers versus nonsmokers and identify the effect of tramadol and nalbuphine between these groups.A comparative cross-Sectional design will be employed from Allama Iqbal Teaching Hospital, DG Khan, over four months. Participants will be stratified into subgroups receiving either tramadol or nalbuphine.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and female patients are included.
* Adults' patients with Greater than 30 years of age
* Both Smoker and non-Smokers patients are added (Patients who are chain smoker at least 10 cigarettes per day).

Exclusion Criteria:

* Patients are excluded if they have smoking history other than cigarettes smoking like Vapes, Cigar and smokeless tobacco.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study anticipates revealing significant variations in pain perception and analgesic requirements, potentially guiding tailored perioperative protocols for smokers. By addressing gaps in pain management strategies specific to smoking status, this research could enhance postoperative recovery outcomes and inform clinical practices for optimizing analgesia in diverse patient populations.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  The Visual Analog Scale (VAS) is a tool used to measure pain intensity, mood, or other subjective experiences. It typically involves a 10 cm (100mm) line with descriptive anchors at each end, such as "no pain" and "worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Allama Iqbal Teaching hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No